CLINICAL TRIAL: NCT00190437
Title: ANTEAB: a Study of Early Antibiotherapy in the ICU Management of Acute Exacerbations of COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Aurémie GUIMFACK, Department Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P010310
Record Dates: First submitted 2005-09-15; First posted 2005-09-19 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2007-03

CONDITIONS: Chronic Obstructive Lung Disease (COLD)
Keywords: Chronic Obstructive Lung Disease (COLD); Randomized Clinical Trial; Antibiotics; Acute Exacerbation; Mechanical; Ventilation; Intensive Care; Length of Stay; Mortality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Amoxicillin-clavulanic
  Interventions: Drug: Amoxicillin-clavulanic

INTERVENTIONS:
Drug: Amoxicillin-clavulanic — Amoxicillin-clavulanic

SUMMARY:
Intensive Care Unit (ICU) admission for acute exacerbation of chronic obstructive lung disease (COLD) is a major cause of morbidity and mortality in such patients. Although bacterial of mortality in such patients. Although bacterial and or viral infections are considered as the major precipitating factor, the antibiotic strategy in this setting is unclear. The absence of overt infection remains controversial, and has not been adequately studied in patients admitted to the ICU. To assess the benefit ( or lack thereof ) of routine early systemic antibiotic therapy in patients with COLD admitted to the ICU.

The primary objective of the essay is to evaluate the effectiveness of the precocious antibiotic therapy on the length of the respiratory symptoms with the admitted patients in polyvalent medical intensive care of chronic obstructive lung disease ( COLD )

DETAILED DESCRIPTION:
This is a multicenter, randomised, double-blind controlled trial, comparing amoxicillin-clavulanic acid administered for 7 days to a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients included are those with documented or suspected COLD, exclusive of other bronchial or lung disease, and admitted for acute exacerbation, in the absence of overt sepsis or broncho-pneumonia, and having no other organ.

Exclusion Criteria:

* Patients recently hospitalised, having received antibiotics since more than 24h, or on long-term steroids will not be included

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2003-08; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
A 20% reduction of the duration of clinical symptoms of exacerbation is expected | during de study
  A 20% reduction of the duration of clinical symptoms of exacerbation is expected

SECONDARY OUTCOMES:
The incidence of documented infection, antibiotic use, the proportion of patients having infection with resistant bacteria | during the study
  The incidence of documented infection, antibiotic use, the proportion of patients having infection with resistant bacteria

CONTACTS AND LOCATIONS:
Overall Officials: Christian BRUN-BUISSON, Pr,MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Hopital Henri Mondor, Créteil, Val de Marne
  - Assistance Publique-Hopitaux de Paris, Paris, Île-de-France Region